CLINICAL TRIAL: NCT05119764
Title: Manual Lymphatic Drainage Before and After Total Knee Replacement, a Single-center Observer-blinded Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moritz Wagner (Other)
Collaborators: Bezirkskrankenhaus St. Johann in Tirol (Other)
Responsible Party: Sponsor-Investigator, Moritz Wagner, Principal Investigator, Dr. med. univ. Moritz Wagner, Bezirkskrankenhaus St. Johann in Tirol
Organization: Bezirkskrankenhaus St. Johann in Tirol (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1466/2020
Record Dates: First submitted 2021-05-12; First posted 2021-11-15 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Total Knee Arthroplasty; Manual Lymphatic Drainage; MLD; Rehabilitation; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with three treatment groups, two intervention groups and one control group
Who Masked: Investigator
Masking Description: Observer/Investigators are unaware of the treatment arm of each patient. Patients cannot be blinded, due to the obvious treatment intervention (manual lymphatic drainage 15 minutes for 5 days).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Standard pre- and postoperative physical therapy without manual lymphatic drainage.
- Manual lymphatic drainage before and after knee replacement (Experimental): Manual lymphatic drainage before and after knee replacement
  Interventions: Procedure: Manual Lymphatic Drainage
- Manual lymphatic drainage after knee replacement (Experimental): Manual lymphatic drainage after knee replacement
  Interventions: Procedure: Manual Lymphatic Drainage

INTERVENTIONS:
Procedure: Manual Lymphatic Drainage — Manual Lymphatic Drainage is a form of physical therapy with the primary goal of accelerating lymphatic drainage.
  In this study, the manual lymphatic drainage is applied by experienced physical therapists 5 days in a row for 30 minutes each; after and/or before the surgery.
  Arms: Manual lymphatic drainage after knee replacement; Manual lymphatic drainage before and after knee replacement

SUMMARY:
The aim of this observer-blinded randomized controlled trial is the evaluation of the influence of manual lymphatic drainage (MLD) on the outcome of patients receiving total knee replacement (TKA).

ELIGIBILITY:
Inclusion Criteria:

* Total Knee Arthroplasty (TKA)

Exclusion Criteria:

* Venous insufficiency
* BMI > 38
* Vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Volume | Change in swelling weeks before the operation to one year after the operation
  The swelling/volume is calculated through measurements of the circumference at 7 distinct points of the leg. The unit is [mm].
Function | Change in ROM weeks before the operation to one year after the operation
  Knee range of motion (ROM), active and passive. The unit is [degrees]
Knee Pain | Change in pain weeks before the operation to one year after the operation
  Visual analogue scale from 0 to 10 on the average level of knee pain in the last 24 hours.

SECONDARY OUTCOMES:
Subjective patient reported outcome | Before the operation, five days after the operation and one year after the operation
  WOMAC Score (Western Ontario and McMaster University Osteoarthritis Index)

CONTACTS AND LOCATIONS:
Locations (1):
- BKH St. Johann in Tirol, Sankt Johann in Tirol, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Undecided